CLINICAL TRIAL: NCT00224107
Title: A Multi-Center, Randomized, Double-Blind, Placebo Controlled, Parallel Evaluation of the Efficacy and Safety of a New Drug in the Treatment of the Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: A New Drug for Benign Prostatic Hyperplasia (BPH) Compared With Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Gary Hoel, RPh, PhD, Executive Director of Clinical Research, Watson Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SI04009
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2009-12-03 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Benign prostatic hyperplasia, BPH, alpha blocker
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — silodosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silodosin (Experimental): Silodosin 8 mg once daily with food
  Interventions: Drug: Silodosin
- placebo (Placebo Comparator): Matching Placebo capsule once daily with food
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Silodosin — 8 mg daily for 12 weeks
  Other Names: Rapaflo
  Arms: Silodosin
Other: Placebo — 1 capsule daily for 12 weeks
  Arms: placebo

SUMMARY:
A new drug for benign prostatic hyperplasia is compared to placebo for to determine if it is safe and effective. The study lasts approximately 20 weeks.

DETAILED DESCRIPTION:
This will be a multi-center, double-blind, placebo controlled, parallel, 12 week treatment trial in men with signs and symptoms of benign prostatic hyperplasia. The following procedures are utilized: physical exams, electrocardiograms, clinical laboratory tests, vital signs, the International Prostate Symptom Score, maximum urine flow rate, pharmacokinetics, adverse events, concomitant medications, quality of life, and compliance.

ELIGIBILITY:
Inclusion Criteria:

* Males in good general health and at least 50 years of age, with symptoms of moderate to severe benign prostatic hyperplasia.

Exclusion Criteria:

* Medical conditions that would confound the efficacy evaluation.
* Medical conditions in which it would be unsafe to use an alpha-blocker.
* The use of concomitant drugs that would confound the efficacy evaluation.
* The use of concomitant drugs that would be unsafe with this alpha-blocker.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2005-05; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hill, PharmD, RPh, Study Director — Watson Pharmaceuticals
Locations (43):
- United States (43):
  - Huntsville, Alabama
  - Tucson, Arizona
  - Anaheim, California
  - Culver City, California
  - Irvine, California
  - La Jolla, California
  - Long Beach, California
  - Newport Beach, California
  - San Diego, California
  - Aurora, Colorado
  - Wheat Ridge, Colorado
  - Waterbury, Connecticut
  - Aventura, Florida
  - Clearwater, Florida
  - Coral Gables, Florida
  - Pensacola, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Des Moines, Iowa
  - Saint Joseph, Michigan
  - Edina, Minnesota
  - Missoula, Montana
  - Las Vegas, Nevada
  - Bay Shore, New York
  - Garden City, New York
  - Manhasset, New York
  - New York, New York
  - Staten Island, New York
  - Williamsville, New York
  - Charlotte, North Carolina
  - Salisbury, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Bethany, Oklahoma
  - Portland, Oregon
  - Lancaster, Pennsylvania
  - Greer, South Carolina
  - Dallas, Texas
  - Salt Lake City, Utah
  - Lakewood, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin

REFERENCES:
- [Result] Marks LS, Gittelman MC, Hill LA, Volinn W, Hoel G. Rapid efficacy of the highly selective alpha1A-adrenoceptor antagonist silodosin in men with signs and symptoms of benign prostatic hyperplasia: pooled results of 2 phase 3 studies. J Urol. 2009 Jun;181(6):2634-40. doi: 10.1016/j.juro.2009.02.034. Epub 2009 Apr 16. PMID 19371887
- [Derived] Marks LS, Gittelman MC, Hill LA, Volinn W, Hoel G. Rapid efficacy of the highly selective alpha(1A)-adrenoceptor antagonist silodosin in men with signs and symptoms of benign prostatic hyperplasia: pooled results of 2 phase 3 studies. J Urol. 2013 Jan;189(1 Suppl):S122-8. doi: 10.1016/j.juro.2012.11.020. PMID 23234617
- [Derived] Roehrborn CG, Kaplan SA, Lepor H, Volinn W. Symptomatic and urodynamic responses in patients with reduced or no seminal emission during silodosin treatment for LUTS and BPH. Prostate Cancer Prostatic Dis. 2011 Jun;14(2):143-8. doi: 10.1038/pcan.2010.46. Epub 2010 Dec 7. PMID 21135869

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Silodosin | Placebo
Started | 233 | 228
Completed | 202 | 214
Not Completed | 31 | 14
Not completed — Adverse Event | 20 | 6
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silodosin | Placebo | Total
Number analyzed (Participants) | 233 | 228 | 461
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 136 | 130 | 266
  >=65 years | 97 | 98 | 195
Age Continuous [Mean (Standard Deviation); unit: years] | 64.4 (7.94) | 64.0 (7.84) | 64.2 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 233 | 228 | 461
Region of Enrollment [Number; unit: participants]
  United States | 233 | 228 | 461

OUTCOME MEASURES:

1. Primary Outcome: International Prostate Symptom Score (IPSS)
Description: Change from baseline In IPSS at Week 12. IPSS uses a 0 to 35 scale; 0 best, 35 worse symptoms
Time Frame: 12 weeks
Population: The number of participants for analysis is determined by Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: Units on a 0 to 35 scale
Arm/Group | Silodosin | Placebo
Number analyzed (Participants) | 233 | 228
Units on a 0 to 35 scale
  Baseline IPSS | 21.5 (5.38) | 21.4 (4.91)
  Change from Baseline in IPSS at Week 12 | -6.5 (6.73) | -3.6 (5.85)

2. Secondary Outcome: Maximum Urine Flow Rate (Qmax)
Description: Change from baseline in maximum urine flow rate (Qmax)at Week 12
Time Frame: 12 weeks
Population: The number of participants for analysis is determined by Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | Silodosin | Placebo
Number analyzed (Participants) | 233 | 228
mL/sec
  Baseline Qmax | 9.0 (2.60) | 9.0 (2.85)
  Change from Baseline in Qmax at Week 12 | 2.2 (4.31) | 1.2 (3.81)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Silodosin | Placebo
Serious Adverse Events (participants affected / at risk) | 3/233 | 3/228
Other Adverse Events (participants affected / at risk) | 116/233 | 24/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silodosin (N=233) | Placebo (N=228)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Silodosin (N=233) | Placebo (N=228)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6) | 4 (4)
Headache (Nervous system disorders) | 8 (8) | 3 (4)
Insomnia (Nervous system disorders) | 5 (5) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 7 (7)
Orthostatic hypotension (Vascular disorders) | 6 (6) | 5 (7)
Retrograde ejaculation (Reproductive system and breast disorders) | 68 (70) | 2 (2)
Sinusitis (Infections and infestations) | 5 (6) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less